CLINICAL TRIAL: NCT00512616
Title: An Investigation of the Efficacy of the Glutamate Transporter GLT 1 in the Treatment of Bipolar Depression
Brief Title: A Glutamate Transporter GLT1, in the Treatment of Bipolar Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Carlos A. Zarate, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070201; 07-M-0201
Record Dates: First submitted 2007-08-04; First posted 2007-08-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-15

CONDITIONS: Bipolar Disorder
Keywords: Ceftriaxone; Acute Antidepressant Effects; Glutamatergic System; Double-Blind; Mood Disorders; Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Ceftriaxone

SUMMARY:
This study examines if Ceftriaxone, an antibiotic, will improve symptoms of depression in Bipolar Disorder.

Purpose: This study will examine whether the drug ceftriaxone can help patients with bipolar depression during short-term treatment of symptoms such as depressed mood, psychomotor retardation (slowed down thinking and movements), and problems with sleep. Recent studies suggest that abnormalities in the brain levels of the chemical glutamate may be involved in causing depression. Ceftriaxone increases a protein in the brain called GLT1, which is responsible for regulating brain levels of glutamate.

People between 18 and 65 years of age with bipolar disorder who are currently in a depressive episode of at least 4 weeks but no longer than 12 months duration may be eligible for this study.

Participants are admitted to the NIH Clinical Center for about 10 weeks. During the first 1 to 2 weeks, they are evaluated and tapered off any antidepressant or mood stabilizers they have been taking. They remain free of all medication for 2 weeks and are then randomly assigned to take either ceftriaxone or placebo for 6 weeks. The study drugs are given intravenously (through a vein) every day. To minimize discomfort, patients are given a PICC line - a tube that is inserted in a vein in the arm and remains there for the duration of drug treatment. This prevents the need for repeated intravenous injections.

Patients have a physical examination at the beginning and at the end of the study and two electrocardiograms (ECG) during the study. They are evaluated periodically with a series of psychiatric rating scales to determine the effects of the study drug on mood and thinking and they have periodic blood tests to assess their health status.

In addition, patients are asked to undergo a lumbar puncture (spinal tap) twice during the study to collect a sample of cerebrospinal fluid (CSF, the fluid that bathes the brain and spinal cord). The CSF is examined to try to understand how brain chemicals are related to depression and to the effects of ceftriaxone. A local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle. This test is optional.

At the end of the study patients are offered free treatment for up to 3 months with standard medications for bipolar depression and a referral to a community physician for long-term treatment will be made.

DETAILED DESCRIPTION:
Bipolar affective disorder (BPD, manic-depressive illness) is a common, severe, chronic and often life-threatening illness. Increasingly, it is being recognized that it is the depressive phase of the illness, which contributes much of the morbidity and mortality. To date, only a few of the available somatic treatments have been proven to be effective for the acute phase of bipolar depression. Thus, there is a clear need to develop novel and improved therapeutics for bipolar depression. Recent preclinical studies suggest that antidepressants may exert delayed indirect effects on the glutamatergic system. Clinical data suggests that glutamatergic modulators may have antidepressant effects in humans. We first tested the glutamatergic modulator riluzole, an inhibitor of glutamate release and enhancer of glutamate reuptake in astrocytes and found it to have antidepressant properties in patients with treatment-resistant major depression and bipolar depression. In a recent study, we found that a single intravenous dose of the non-competitive NMDA antagonist ketamine produced a rapid and relatively sustained antidepressant effect in patients with treatment-resistant major depression. A recent report found that the Beta-lactam antibiotic ceftriaxone increased uptake of glutamate via increased GLT1 function (Rothstein et al 2005) and had antidepressant-like effects in animal models (Mineur et al 2006). Together, these data suggest that the glutamatergic system may play a role in the pathophysiology and treatment of depression, and that agents which more directly reduce glutamatergic neurotransmission may represent a novel class of antidepressants.

We propose to expand our previous findings on the efficacy of glutamatergic modulators in patients with unipolar and bipolar depression by testing a specific, new mechanism where by we use ceftriaxone to chronically increase the expression of the glutamate transporter GLT1 in order to facilitate the removal of glutamate from the synaptic cleft in an effort to reduce excessive glutamate transmission and as a result produce acute antidepressant effects. The model presented here is a clinical testable one, and one that, if successful, holds the potential to develop a group of novel pharmacological treatments for major depression.

Patients, ages 18 to 65, with a diagnosis of bipolar depression (without psychotic features), will be randomized to double-blind treatment to receive either ceftriaxone (1-4 g/day) or placebo intravenously for a period of 6 weeks. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria. Approximately 86 patients with bipolar depression will be enrolled in the study.

ELIGIBILITY:
* INCLUSION CRITERIA

Male or female subjects, 18 to 65 years of age.

Female subjects of childbearing potential must be using a medically accepted means of contraception.

Each subject must have a level of understanding sufficient to agree to all required tests and examinations.

Each subject must understand the nature of the study and must sign an informed consent document.

Subjects must fulfill the criteria for bipolar I or II disorder, current episode depressed without psychotic features as defined in DSM-IV based on clinical assessment and confirmed by structured diagnostic interview SCID-P.

Subjects must have an initial score at Visit 1 and Visit 2 of at least 20 on the MADRS.

Subjects must have an initial score at Visit 1 and Visit 2 of less than or equal to 12 on the YMRS.

Current duration of depressive episode should be at least 4 weeks (full criteria) but no longer than 12 months in duration.

For Bipolar II, subjects must have experienced, in the opinion of the investigator, at least two previous hypomanic and two major depressive episodes as defined in DSM-IV.

EXCLUSION CRITERIA

Presence of psychotic features.

Female subjects who are either pregnant or nursing.

Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Current or past colitis.

Subjects with uncorrected hypothyroidism or hyperthyroidism.

Clinically significant abnormal laboratory tests.

Current or past blood dyscrasia.

Documented history of hypersensitivity or intolerance to penicillins, cephalosporins or ceftriaxone.

Subjects who are immunocompromised.

DSM-IV substance abuse or dependence within the past 90 days.

Current or past seizure disorder.

Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to Visit 2.

Treatment with a reversible MAOI, guanethidine, or guanadrel within 1 week or with fluoxetine within 5 weeks prior to Visit 2.

Treatment with any other concomitant medication with primarily CNS activity, other than specified in Appendix A of the protocol.

Treatment with clozapine or ECT within 4 weeks prior to Visit 2.

Current diagnosis of schizophrenia or other psychotic disorder as defined in the DSM-IV.

Diagnosed with an axis I disorder other than bipolar disorder that was the primary focus of treatment within 6 months before the screening.

MADRS score of greater than 4 on item 10 (active suicidal plan).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08-01; Primary Completion 2009-09-15 (Actual); Study Completion 2009-09-15 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of acute ceftriaxone therapy compared with placebo in pts with bipolar disorder current episode depressed w/o psychotic features, in improving overall depressive symptomatology. | 6-weeks

SECONDARY OUTCOMES:
Assess the efficacy of acute ceftriaxone therapy compared with placebo in pts with bipolar disorder current episode depressed w/o psychotic features, in improving overall depressive symptomatology. | 6-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bannerman DM, Good MA, Butcher SP, Ramsay M, Morris RG. Distinct components of spatial learning revealed by prior training and NMDA receptor blockade. Nature. 1995 Nov 9;378(6553):182-6. doi: 10.1038/378182a0. PMID 7477320
- [Background] Benoit E, Escande D. Riluzole specifically blocks inactivated Na channels in myelinated nerve fibre. Pflugers Arch. 1991 Dec;419(6):603-9. doi: 10.1007/BF00370302. PMID 1664937
- [Background] Bittner MJ, Dworzack DL, Preheim LC, Tofte RW, Crossley KB. Ceftriaxone therapy of serious bacterial infections in adults. Antimicrob Agents Chemother. 1983 Feb;23(2):261-6. doi: 10.1128/AAC.23.2.261. PMID 6301365